CLINICAL TRIAL: NCT05357703
Title: Evaluation of the Efficacy of a Home-Use Photobiomodulation Device for the Treatment of Patients With Knee Osteoarthritis: An Open Label, Single-Arm Clinical Trial
Brief Title: Efficacy of a Home-Use Photobiomodulation Device for the Treatment of Patients With Knee Osteoarthritis
Acronym: PBM&KOA-02
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erika Carmel ltd (Other)
Collaborators: Holy Family Hospital, Nazareth, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFH-256-2022
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
Keywords: Photobiomodulation; Low-Level Laser Therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard treatment + Active B-Cure laser (Experimental): Subjects from Standard treatment + Active B-Cure laser will receive standard care and in addition will self-treat at home with the B-Cure device.
  Interventions: Device: Standard treatment + Active B-Cure laser

INTERVENTIONS:
Device: Standard treatment + Active B-Cure laser — The B-Cure laser pro is a portal, non-invasive, photobiomodulation device, that emits light in the near infrared (808nm) over an area of 1X4.5 cm2 with power output of 250mW, and energy dose of 5J/minute.

SUMMARY:
Osteoarthritis is a degenerative disease affecting joint cartilage and its surrounding tissue. It is the leading cause of disability in the elderly. Photobiomodulation (PBM), has been used widely for alleviation of pain, reduction of inflammation, and acceleration of wound healing, and particularly to treat knee osteoarthritis (KOA). The purpose of the current study is to determine if B-Cure laser treatments, applied at home, by the patient or personal caregiver in a real-life situation, can reduce pain and improve functionality in patients with KOA.

DETAILED DESCRIPTION:
Eligible patients with knee osteoarthritis will receive a B-Cure laser device for self-application at home in addition to standard care. Patients will be invited to the clinic for 3 visits: baseline, 1, and 2 months. Evaluations at the visits will include physical examination, knee range of motion, time up&go test, and patient reported outcomes including subjective pain level by visual analogue scale (VAS), functional and quality of life questionnaires.

The study hypothesis is that B-Cure laser treatments, applied, at home, by the patient, can ameliorate KOA related inflammation thereby reducing pain and improving functionality in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnoses of knee osteoarthritis by American College of Rheumatology (ACR)
2. Kellgren & Lawrence classification 2-3
3. Knee pain on movement 40 to 90 mm Visual Analog Scale
4. Knee pain and related functional reduction for the last ≥ 3 months
5. Agrees not to use NSAIDs throughout the experiment

Exclusion Criteria:

1. Pregnant or nursing, or with the ability to become pregnant and not using an accepted form of birth control
2. Other causes of knee-related pain (e.g. hip OA, arterial insufficiency, radiculopathy etc) have been ruled out by physical examinations.
3. Knee surgery for KOA
4. Intra-articular steroid injection and/or oral steroid treatment within the last six months
5. Rheumatoid arthritis
6. Active malignancy
7. Uncontrolled diabetes mellitus
8. Neurological conditions: sciatica, neuropathy, multiple sclerosis
9. Other chronic pain conditions that may affect results: Fibromyalgia, back pain, hip pain
10. Has any photobiomodulation (low level laser) device at home or has previously used photobiomodulation for knee pain
11. Has known dermatological sensitivity to light
12. Enrolled in any other clinical trial within the last 6 weeks or enrollment in another clinical trial during participation in this trial.

    -

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-26 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
level of pain | one month
  Change from baseline in pain score by VAS

SECONDARY OUTCOMES:
Change from baseline in WOMAC score [ time point - 1 month] | one month
  The WOMAC is a disease-specific tool used for people with hip or knee OA to measure physical function, pain, and stiffness. It widely used in clinical studies as primary or secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Hadad, MD, Principal Investigator — The Holy Family Hospital, Nazareth, Israel
Locations (1):
- Holy Family Hospital, Nazareth, Israel